CLINICAL TRIAL: NCT05086692
Title: A Phase 1/2 Open Label, Dose Escalation and Expansion Study of MDNA11, IL-2 Superkine, Administered Alone or in Combination With Immune Checkpoint Inhibitor in Patients With Advanced Solid Tumors
Brief Title: A Beta-only IL-2 ImmunoTherapY Study
Acronym: ABILITY-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medicenna Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MDNA11-01; KEYNOTE-E53 (Other: Merck Sharp & Dohme, LLC); MK3475-E53 (Other: Merck Sharp & Dohme, LLC); 2023-507536-21-00 (EU CTIS Number)
Record Dates: First submitted 2021-09-10; First posted 2021-10-21 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor; Unresectable Solid Tumor; Clear Cell Renal Cell Carcinoma; Triple Negative Breast Cancer; Non-Small Cell Lung Cancer Squamous; Non-Small Cell Lung Cancer Non-squamous; Colorectal Cancer (MSI-H); Gastric Cancer; Cervical Cancer; Basal Cell Carcinoma; Bladder Cancer; Merkel Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Cutaneous Squamous Cell Carcinoma; Pleural Mesothelioma; Esophageal Cancer; Endometrial Carcinoma; Solid Tumor; Solid Tumor, Adult; MSI-H Solid Malignant Tumor; Cancer With A High Tumor Mutational Burden; Epithelial Ovarian Carcinoma; Primary Peritoneal Cancer; Gastroesophageal Junction (GEJ) Cancer; Acral Melanoma; Mucosal Melanoma; Cutaneous Melanoma; DMMR Solid Malignant Tumor; Fallopian Tube Cancer; Ovarian Cancer; MSI-H Cancer; DMMR Cancer; Pancreas Adenocarcinoma (MSI-H); Skin Cancer; Viral Cancer; Cervical Cancers; Endometrial Cancer
Keywords: IL-2; IL2; Interleukin-2; cancer; metastatic; ccRCC; TNBC; NSCLC; CRC; GEJ; intrahepatic; extrahepatic; MCC; SCCHN; CSCC; Gastroesophageal Junction; advanced; unresectable; MSI-H; dMMR; Microsatellite Instability-High; Mismatch Repair Deficient; PD-1; immunotherapy; anti-PD-1; BCC; RCC; HCC; Tumor Mutation Burden High; TMB-H; PDAC
MeSH Terms: conditions — Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Basal Cell; Urinary Bladder Neoplasms; Carcinoma, Merkel Cell; Squamous Cell Carcinoma of Head and Neck; Mesothelioma, Malignant; Esophageal Neoplasms; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial; Neoplasms; Melanoma; Fallopian Tube Neoplasms; Ovarian Neoplasms; Skin Neoplasms; Neoplasm Metastasis; Turcot syndrome | interventions — Interleukin-2; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation (MDNA11 monotherapy and MDNA11 + pembrolizumab) followed by dose expansion with MDNA11 monotherapy and combination (MDNA11 + pembrolizumab).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MDNA11 (Experimental): MDNA11 is a long-acting "beta-only" recombinant interleukin-2 (rIL-2) albumin fusion
  Interventions: Drug: MDNA11; Drug: Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: MDNA11 — MDNA11 will be administered, IV on a once every 2 weeks (Q2W) dosing schedule. Provisional dose cohorts for monotherapy dose escalation doses ranging from 0.003 to 0.6 (mg/kg): until determining the monotherapy Recommended Dose for Expansion (mRDE).
  Other Names: Interleukin-2 (IL-2)-albumin
Drug: Pembrolizumab (KEYTRUDA®) — MDNA11 will be administered in combination with pembrolizumab, IV. MDNA11 dose range to be evaluated in combination with pembrolizumab until determining the combination Recommended Dose for Expansion (cRDE).

SUMMARY:
This is a Phase 1/2, multi-center, open-label, dose-escalation and expansion study to evaluate safety and tolerability, PK, pharmacodynamic, and early signal of anti-tumor activity of MDNA11 alone or in combination with a checkpoint inhibitor in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study drug, MDNA11, long-acting "beta-only" recombinant interleukin-2 (rIL-2). MDNA11 specifically engineered to overcome the shortcomings of rhIL-2 (aldesleukin) by preferentially activating immune effector cells (CD8+ T- and NK cells) responsible for killing cancer cells, with minimal or no stimulation of immunosuppressive Tregs. It is designed to potentially enhance host immune response and fusion to albumin increases the half-life further avoiding frequent dosing required with rhIL-2.

The study will be conducted at up to 30 clinical sites following regulatory authority and institutional review board / independent ethics committee (IRB/ IEC) approval and completion of informed consent. The study will be conducted in multiple parts:

* Monotherapy (MDNA11 alone) dose escalation
* Monotherapy (MDNA11 alone) dose expansion in select tumor types
* Combination (MDNA11 + pembrolizumab) dose escalation
* Combination (MDNA11 + pembrolizumab) dose expansion in select tumor types

Approximately 115 patients will be enrolled.

After commencing treatment (first exposure of MDNA11 alone or MDNA11 + pembrolizumab), tumor assessment by CT/MRI will be performed every 8 weeks ± 1 week until immune confirmed progressive disease ("iCPD") by iRECIST, discontinuation of study drug(s), withdrawal of consent or loss to follow-up. Treatment beyond progression may be permitted if criteria are met. Patients can withdraw from participation at any time.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged at least 18 years (inclusive at the time of informed consent).
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
3. Must be able and willing to provide written informed consent prior to start of any study procedures and assessments and must be willing to comply with all study procedures.
4. Histologically or cytologically confirmed locally advanced or metastatic solid tumor (see tumor types listed under conditions)
5. Demonstrated adequate organ function
6. Measurable disease as per Response Evaluation Criteria in Solid Tumors, (RECIST v1.1) and documented by CT and/or MRI.
7. Life expectancy of ≥ 12 weeks.
8. Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening and within 72 hours before the first dose of study drug(s). Women must not be breastfeeding.
9. Agree to use highly effective contraception methods. WOCBP must agree to use highly effective birth control.

Key Exclusion Criteria:

1. Last administration of prior antitumor therapy:

   * Prior systemic anti-cancer therapy including investigational agents within 4 weeks (could consider shorter interval for kinase inhibitors or other short half-life drugs) prior to start of treatment.
   * Prior radiotherapy within 2 weeks prior to start of treatment or has had a history of radiation pneumonitis. A 1-week washout is required for palliative radiation (<2 weeks of radiotherapy) to non-CNS disease.
   * Radiation therapy to the lung that is > 30Gy within 6 months prior to start of treatment.
   * Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to start of treatment. Concomitant participation in an observational study must be discussed on a case-by-case basis with the MM for approval.
2. Has known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to start of treatment, subject to discussion with MM.
3. Active malignancy (other than the disease under treatment in the study) within the previous 3 years except for curable cancers.
4. Condition requiring long-term systemic treatment with either corticosteroids > 10 mg daily prednisone equivalent or any other form of immunosuppressive therapy within 7 days prior to start of treatment.
5. Clinically significant active, known or suspected autoimmune disease, or diseases that can be exacerbated with immunotherapy.
6. Severe pulmonary, cardiac or other systemic disease.
7. Known hepatitis B or C virus infection.
8. Females who are pregnant or lactating or planning to become pregnant during the study.
9. Has had an allogeneic tissue/solid organ transplant.
10. Active infection requiring systemic therapy.
11. Any medical, emotional or psychiatric condition that interfere with the patient's ability to adhere to the protocol
12. Any other underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug(s) unsafe or obscure the interpretation of toxicity determination or adverse events.
13. Known severe hypersensitivity to any component of study drug(s).
14. Inability to comply with study and follow up procedures as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male Female (Women of Childbearing Potential will be subject to pregnancy testing)
Enrollment: 115 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
MDNA11 Recommended Dose for Expansion for monotherapy (mRDE) and Recommended Dose for Expansion for combination (cRDE) | 24 months
  Evaluation of tolerability as measured by number of patients with dose limiting toxicities (DLTs)
Incidence of Treatment Related Adverse Events (TRAEs) | 24 months
  Rate of TRAEs in patients with advanced solid tumors
Incidence of Treatment Emergent Adverse Events (TEAEs) | 24 months
  Rate of TEAEs in patients with advanced solid tumors

SECONDARY OUTCOMES:
Pharmacokinetic characteristics on MDNA11 - Cmax (ug/mL) | Up to 24 months
  Maximum observed serum drug concentration
Pharmacokinetic characteristics on MDNA11 - Tmax (h) | Up to 24 months
  Time to maximum observed serum drug concentration
Pharmacokinetic characteristics on MDNA11 - AUClast (h.ug/mL) | Up to 24 months
  Area under the serum concentration vs time curve from time zero to the last measurable concentration
Immunogenicity of MDNA11 (anti-drug antibodies) | Up to 24 months
  Incidence and persistence of anti-drug antibodies to MDNA11
Pharmacodynamic effects of MDNA11 | Up to 24 months
  Measurement of translational parameters - Flow cytometry analysis of immune cells in blood and serum measurements of cytokine levels
Anti-tumor activity of MDNA11 (alone or in combination with CPI) - Overall Response Rate (ORR) | Approximately 24 months
  Assessed by RECIST v1.1 and iRECIST; CR+PR/Evaluable N
Anti-tumor activity of MDNA11 (alone or in combination with CPI) - Disease Control Rate (DCR) | Approximately 24 months
  CR+PR+SD/Evaluable N
Anti-tumor activity of MDNA11 (alone or in combination with CPI) - Progression Free Survival (PFS) | Approximately 24 months
  Time from signing ICF to disease progression

OTHER OUTCOMES:
Analysis of immune characteristics of the tumor microenvironment | Up to 24 months
  Measured by change in Tumor Infiltrating Lymphocyte (TIL) levels

CONTACTS AND LOCATIONS:
Overall Officials: Nina Merchant, Study Director — Medicenna Therapeutics; Arash Yavari, MBBS, Study Chair — Medicenna Therapeutics
Locations (27):
- United States (7):
  - Sharp Memorial Hospital, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Emory - Winship Cancer Institute, Atlanta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Scientia Clinical Research, Randwick, New South Wales
  - Macquarie University, Sydney, New South Wales
  - University of the Sunshine Coast, Buderim, Queensland
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Mater Misericordiae University Hospital, Dublin, Ireland
- Portugal (2):
  - START Lisbon - Centro de Ensaios Clínicos, ULS Sta Maria, Lisbon
  - Instituto Portugues De Oncologia Do Porto, Porto
- South Korea (4):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea St. Vincent Hospital, Suwon, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu
- Spain (8):
  - Institut Catala d'Oncologia (ICO)-Badalona, Badalona
  - START Barcelona / HM Nou Delfos, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - START Madrid / Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Hospital Universitario de Torrejon, Torrejón

IPD SHARING:
Plan to Share IPD: No